CLINICAL TRIAL: NCT02732197
Title: Effects of Sedation on Spinal Anesthesia-induced Maternal Hypotension in Preoperatively Anxious Parturients Undergoing Urgent Category-1 Cesarean Section: A Historical Cohort Study
Brief Title: Effects of Sedation on Spinal Anesthesia-induced Maternal Hypotension
Status: Completed | Type: Observational
Sponsor: Van Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr.Cenk Sahan, Attending Anesthesiologist, Van Training and Research Hospital
Other Study IDs: 2015/4
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Cesarean Section; Preoperative Anxiety; Spinal Anesthesia; Sedation; Maternal Hypotension
MeSH Terms: interventions — Thiopental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sedation (S): Parturients who received IV thiopental 2 mg kg-1 and if necessary additional 50 mg immediately after spinal anesthesia until reaching at least Ramsay sedation score of 3 (1: patient anxious, agitated or restless, 6: patient with no response to light glabella tap or loud auditory stimulus.).
  Interventions: Drug: Sedation
- No sedation (NS): Parturients who did not receive any sedative agent after the spinal anesthesia performance.
  Interventions: Drug: No sedation

INTERVENTIONS:
Drug: Sedation — Parturients who received IV thiopental 2 mg kg-1 and if necessary additional 50 mg immediately after spinal anesthesia until reaching at least Ramsay sedation score of 3 (1: patient anxious, agitated or restless, 6: patient with no response to light glabella tap or loud auditory stimulus.).
  Other Names: Thiopental
  Groups: Sedation (S)
Drug: No sedation — Parturients did not receive any type of sedation after spinal anesthesia.
  Other Names: No drug
  Groups: No sedation (NS)

SUMMARY:
Background: This study was designed to investigate the effect of sedation on the occurrence of maternal hypotension in preoperatively anxious parturients undergoing urgent category-1 Cesarean section (C/S) under spinal anesthesia.

Methods: After institutional ethics committee approval, prospectively collected data of 1824 parturients undergoing C/S were reviewed. Parturients with high preoperative anxiety scores (visual analogue scale for anxiety (VAS-A)≥70) undergoing C/S under spinal anesthesia with thiopental (Group S=49) and without any other type of sedation (Group NS=53) were included in the analysis. Hemodynamic parameters were documented and maximum systolic arterial pressure (SAP) reductions from the baseline after spinal anesthesia were calculated. Incidences of hypotension (SAP≥30% decrease from baseline or <100 mmHg) and bradycardia (HR<55 beats/min), and related-ephedrine and -atropine requirements were noted. Our primary endpoint was to compare the maximum SAP reductions from the baseline values in Groups S and NS. Secondary endpoints were incidences of hypotension and bradycardia, required ephedrine and atropine doses, newborn Apgar scores at 1st and 5th min.

DETAILED DESCRIPTION:
Background: This study was designed to investigate the effect of thiopental sodium sedation on the occurrence of maternal hypotension in preoperatively anxious parturients undergoing urgent category-1 Cesarean section (C/S) under spinal anesthesia.

Methods: After institutional ethics committee approval, prospectively collected data of 1824 parturients undergoing C/S at Van Training and Research Hospital between August 2014 and February 2015 were reviewed. Parturients with high preoperative anxiety scores (visual analogue scale for anxiety (VAS-A)≥70) undergoing C/S under spinal anesthesia with thiopental (Group S=49) and without any other type of sedation (Group NS=53) were included in the analysis. All parturients received SA with hyperbaric bupivacaine 0.5% 2.5 mL. Hemodynamic parameters were documented and maximum systolic arterial pressure (SAP) reductions from the baseline after spinal anesthesia were calculated. Incidences of hypotension (SAP≥30% decrease from baseline or <100 mmHg) and bradycardia (HR<55 beats/min), and related-ephedrine and -atropine requirements were noted. All data were obtained from the surgical database and patient charts. Primary endpoint of our study was to compare the maximum SAP reductions from the baseline values in Groups S and NS. Secondary endpoints were incidences of hypotension and bradycardia, required ephedrine and atropine doses, newborn Apgar scores at 1st and 5th min.

ELIGIBILITY:
Inclusion Criteria:

* Urgent category-1 C/S
* ASA physical status I-II
* Aged between 18 and 35 years
* Term (≥37 weeks) singleton pregnancy
* BMI <40 kg/m2
* Height >150 cm or <180 cm
* High preoperative anxiety scores (visual analogue scale for anxiety (VAS-A) ≥70)
* Spinal anesthesia with thiopental sodium sedation
* Spinal anesthesia without any sedation

Exclusion Criteria:

* Preoperative prehydration
* Placenta previa
* Placenta accreta
* Hypertension
* Pregnancy-induced hypertension
* Urgent category ≥2
* General anesthesia
* Spinal anesthesia with sedation other than thiopental sodium

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Parturients undergoing urgent category-1 Cesarean section (C/S) under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Maximum systolic arterial pressure (SAP) reductions from the baseline values | 0-10 minutes
  % SAP reduction after spinal anesthesia

SECONDARY OUTCOMES:
Incidence of maternal hypotension | 0-30 minutes
  Incidence of hypotension during the surgery (decrease in SAP >30% from baseline or an absolute value <100 mmHg)
Incidence of maternal bradycardia | 0-30 minutes
  Incidence of bradycardia during the surgery (heart rate (HR) <55 beats min-1)
Ephedrine requirement | 0-30 minutes
  Ephedrine 5 mg IV boluses were administered with 2 min intervals until SAP returned to a value of >100 mmHg
Atropine requirement | 0-30 minutes
  Bolus of IV 0.5 mg atropine was given if bradycardia (HR <55 beats min-1) occurred
Incidence of maternal nausea | 0-30 minutes
  If any during the Cesarean section, recorded
Incidence of maternal vomiting | 0-30 minutes
  If any during the Cesarean section, recorded
Newborn Apgar score 1st min | 1st min
  Apgar score at 1st min (0-3: severely depressed, 4-6: moderately depressed, 7-10: excellent condition)
Newborn Apgar score 5th min | 5th min
  Apgar score at 5th min (0-3: severely depressed, 4-6: moderately depressed, 7-10: excellent condition)

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Sahan, MD, Principal Investigator — Design and conduct the study, review and analyze the data, and write the manuscript
Locations (1):
- Van Training and Research Hospital, Department of Anesthesiology, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Orbach-Zinger S, Ginosar Y, Elliston J, Fadon C, Abu-Lil M, Raz A, Goshen-Gottstein Y, Eidelman LA. Influence of preoperative anxiety on hypotension after spinal anaesthesia in women undergoing Caesarean delivery. Br J Anaesth. 2012 Dec;109(6):943-9. doi: 10.1093/bja/aes313. Epub 2012 Sep 10. PMID 22964265